CLINICAL TRIAL: NCT03348137
Title: ORIEN-PROGENY Family History Questionnaire Study: Recognizing Inherited Susceptibility to Cancer
Brief Title: Oncology Research Information Exchange Network in Improving Genetic Screening Rate in Patients With Cancer
Status: Withdrawn | Type: Observational
Why Stopped: PI left
Sponsor: University of Southern California (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 0S-16-16; NCI-2017-01450 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 0S-16-16 (Other: USC / Norris Comprehensive Cancer Center); P30CA014089 (NIH)
Record Dates: First submitted 2017-11-04; First posted 2017-11-20 (Actual); Last update posted 2019-10-24 (Actual); Status verified 2019-10

CONDITIONS: Malignant Neoplasm
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Ancillary-Correlative (questionnaire): Patients take Progeny Genetic Pedigree and Family History Questionnaire. Results are reviewed by the site specific research coordinator and/or genetic counselor to assess whether a patient fulfills criteria for referral to the site specific cancer genetics clinic for further evaluation.
  Interventions: Other: Questionnaire Administration

INTERVENTIONS:
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This research trial studies how well Oncology Research Information Exchange Network (ORIEN) works in improving genetic screening rate in patients with cancer. Implementation of Progeny Genetic Pedigree and Family History Questionnaire software across all ORIEN member institutions may add value and utility for recognizing and caring for patients with an inherited susceptibility to cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Measure the change in uptake of cancer genetic referrals and genetic testing in the ORIEN system of cancer centers implementing the Progeny Family History Questionnaire (FHQ).

SECONDARY OBJECTIVES:

I. Follow and estimate utilization of preventive health behaviors among Progeny FHQ users across all institutions.

II. Compare utilization of preventive health behavior between Progeny FHQ risk identification and genetic testing.

OUTLINE:

Patients take Progeny Genetic Pedigree and Family History Questionnaire. Results are reviewed by the site specific research coordinator and/or genetic counselor to assess whether a patient fulfills criteria for referral to the site specific cancer genetics clinic for further evaluation.

After completion of study, patients are followed up at 6 months after disclosure of genetic testing results.

ELIGIBILITY:
Inclusion Criteria:

* Limited to those patients who are consented to the Total Cancer Care Protocol (TCCP) protocol
* Able to understand and sign the TCCP informed consent, California subject?s bill of rights, Health Insurance Portability and Accountability Act (HIPAA), and research authorization form directly or through an authorized representative; the informed consent, subject?s bill of rights, HIPAA, and research authorization will be available in both English and Spanish languages

Exclusion Criteria:

* Individuals who are not registered as patients for outpatient or inpatient care to the TCCP protocol
* Individuals who are unable to understand or sign the TCCP informed consent, subject?s bill of rights, HIPAA, and research authorization in either English or Spanish

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients consented to the Total Cancer Care Protocol protocol
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2019-07-01 (Estimated); Primary Completion 2037-07-01 (Estimated); Study Completion 2038-07-01 (Estimated)

PRIMARY OUTCOMES:
Changes in Rates of Genetic Testing | Up to 30 months
  Will compare rates of genetic testing before and after implementation of Progeny Family History Questionnaire (FHQ) using the stratified Chi-square test.

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Idos, MD, Principal Investigator — University of Southern California
Locations (1):
- USC / Norris Comprehensive Cancer Center, Los Angeles, California, United States